CLINICAL TRIAL: NCT05317377
Title: Leap Motion Controller Based Exergame Therapy in Geriatric Individuals
Brief Title: Leap Motion In Geriatric Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Farzin Hajebrahimi, PhD, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LeapGeriatric2021
Record Dates: First submitted 2022-03-14; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Elderly
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will be included in the study and randomly divided into two groups using block randomization in Microsoft Excel 'RAND(WS)' function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Exercise (Active Comparator): Structured hand exercises will be applied in 45-minute sessions (16 sessions total), 2 days a week, over 8 weeks in addition to participants' routine physical activities.
  Interventions: Other: Exercise Therapy
- Leap Motion Based Exergame (LMBE) (Experimental): "ErgoActive" and "HandROM" exercise apps focusing on hand exercises and fine motor skills will be applied in 45-minute session (16 sessions total), 2 days a week, over 8 weeks in addition to participants' routine physical activities.
  Interventions: Device: Leap Motion Based Exergame

INTERVENTIONS:
Other: Exercise Therapy — Structured exercises focused on hand functionality
  Arms: Structured Exercise
Device: Leap Motion Based Exergame — Appropriate games from Leap Motion Based Exergame system focused on hand functionality
  Arms: Leap Motion Based Exergame (LMBE)

SUMMARY:
Little is Known about the effects of leap motion based exergame therapy on different functions of elderly adults. The purpose of this study was to evaluate the effect of leap motion based exergame therapy on hand function, cognitive function and quality of life in older adults

ELIGIBILITY:
Inclusion Criteria:

* 50 years old and over,
* having adequate hand function,
* ability to follow commands,
* 24< points in MMSE

Exclusion Criteria:

* presence of exercise contraindications
* 14 or more points on the Geriatric Depression Scale
* diagnosis of dementia
* recent (acute) hand or arm injury

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Grip Strength Test | changes after 8 weeks
  A hand dynamometer (pinch meter gauge; Jamar® Hand Dynamometer - Hydraulic - 200 lb Capacity. Patterson Medical Illinois, USA) will be used to determine the grip strength of the participants. While taking the measurements, the patients will be seated with the shoulder adducted and neutrally rotated, elbow flexed at 90°, forearm and wrist in neutral position. Each grip test will be repeated three times and the highest score for the affected extremity will be used for further analysis.

SECONDARY OUTCOMES:
Pittsburgh Rehabilitation Participation Scale | changes after 8 weeks
  It is a clinician-evaluated outcome scale that examines the patient's participation in therapy and motivation. While the test period lasts 5 minutes, it consists of 6 different scores (1-none/6-excellent). Higher scores mean better performance.
World Health Organization Quality of Life Instrument-Older Adults Module | changes after 8 weeks
  It is a versatile scale that helps to evaluate the quality of life in elderly individuals. WHOQOL-OLD consists of 6 sections: sensory skills, autonomy, past-present-future activities, social participation, death and relationships, and includes 4 items in each section, consisting of a total of 24 questions.
Digit Span Test | changes after 8 weeks
  It consists of two sub-categories, forward and backward number range, and evaluates attention . During the test, the participant is asked to repeat the numbers from 1 to 9 in mixed order, starting from 4 and increasing to 8. At this time, it is important to note that each number is said in one second, slowing down may develop different strategies. The forward range consists of 5 to 7 numbers, while the reverse range consists of 3 to 7 numbers. The participant is asked to count forward or backward from the number said. As many points as they can say are noted as a score.
Duruöz Hand Index | changes after 8 weeks
  It is an 18-item, self-answered scale that evaluates hand activity limitations and its effect on activities of daily living. In the scale where scores between 0-90 can be obtained, high scores indicate low function.
Stroop Test | changes after 8 weeks
  The Stroop Test measures the processing speed, the ability to suppress habitual behavior, focused attention, the ability to do unusual behavior, the ability to change the perceptual setup according to changing demands, and under a disturbing effect. The tests proved to be reliable (with test/retest reliabilities ranging from acceptable (r=0.63) to high (r=0.88) and sensitive to detect small differences in subjects from different age categories.
Purdue Pegboard Test | changes after 8 weeks
  The Purdue Pegboard consists of a board with holes into which metal pegs are inserted by the patient. It also comes with washers and collars to be placed on the pins. The test measures movements, coordination and speed of hand and finger dexterity. In the test procedures, the patient is first asked to use the right hand to properly insert as many pins as possible in the holes. Then, the same procedure is repeated for the left hand. In the final stage the patient is given 60 sec to place the pins, washers and collars using both hands.
Box and Block Test | changes after 8 weeks
  It examines unilateral gross motor skills. A stopwatch, a wooden box with a middle section, and 150 wooden cubes are the required materials. The total duration of the test is 2-5 minutes. The test can be applied between the ages of 6 and 65. Within 60 seconds, which is kept by the stopwatch, it is requested to pass the cubes one by one from one compartment to the other and the number of cubes is noted. This test is applied separately for both extremities.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on reasonable request from the principle investigator. The data are not publicly available due to ethical issues.